CLINICAL TRIAL: NCT01579032
Title: Pulse Wave Analysis and Velocity in Patients With Chronic Renal Failure: a Cross-sectional Observational Study to Assess Association With Left Ventricular Hypertrophy, Uremic Toxins and Inflammation.
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: ML2863
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Arterial Stiffness; CHRONIC RENAL FAILURE; Left Ventricular Hypertrophy
Keywords: CKD,
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CKD patients

SUMMARY:
The aims of the presented study are as follows:

1. To evaluate the endothelial function and arterial stiffness in a large cohort of prevalent CKD patients by means of non-invasive applantion tonometry.
2. To evaluate the association between the serum levels of the representatives of the various classes of uremic toxins and markers of endothelial function and arterial stiffness.
3. To evaluate the association between markers of inflammation and oxidative stress and markers of endothelial function and arterial stiffness.
4. To evaluate the association between echocardiographic parameters and markers of arterial stiffness

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60
* Chronic kidney disease: according to the K-DOQI guidelines ( kidney damage ≥ three months, as defined by structural or functional abnormalities of the kidney, with or without decreased GFR, manifest by either: pathological abnormalities; or markers of kidney damage, including damage in the composition of blood or urine test, or abnormalities in imaging tests; GFR< 60 ml/min/1.73m² for ≥ three months, with or without kidney damage)
* Written informed consent

Exclusion Criteria:

* major illnesses( life expectancy of < 1 year)
* history of atrial fibrillation
* history of myocardial infarction, unstable angina, congestive heart failure, peripheral vascular diasease ,cerebrovascular disease, diabetes

(nonechogenic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CKD patients
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2004-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - University Hospitals, Leuven
  - UZ Leuven, Leuven